CLINICAL TRIAL: NCT06173232
Title: Assessment of Retinal Fundus Imaging Camera
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Digital Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-CLN-001
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Radionuclide Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group 1: Subjects with ETDRS ≥ 35 with or without DME
  Interventions: Device: Camera Imaging
- Group 2: Subjects with ETDRS 20 or less and no DME
  Interventions: Device: Camera Imaging

INTERVENTIONS:
Device: Camera Imaging — Camera Imaging

SUMMARY:
The goal of this prospective study is to evaluate device performance when using fundus images taken from retinal fundus cameras in subjects with and without diabetic retinopathy per ETDRS level 35 and higher with or without macular edema.

DETAILED DESCRIPTION:
The goal of this prospective study is to evaluate device performance when using fundus images taken from retinal fundus cameras in subjects with and without diabetic retinopathy (ETDRS level 35 and higher) with or without macular edema. Study subjects will sign the informed consent form, and data collection will involve being imaged by cameras.

ELIGIBILITY:
Inclusion Criteria:

* 22 years of age or older.
* Documented diagnosis of diabetes mellitus, as per any of the following: Having met the criteria established by the World Health Organization (WHO) and/or the American Diabetes Association (ADA), Hemoglobin A1c (HbA1c) ≥ 6.5%, Fasting Plasma Glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L), Oral Glucose Tolerance Test (OGTT) with two-hour plasma glucose (2-hr PG) ≥ 200 mg/dL (11.1 mmol/L), using the equivalent of an oral 75g anhydrous glucose dose dissolved in water, Symptoms of hyperglycemia or hyperglycemic crisis with a random plasma glucose (RPG) ≥ 200 mg/dL (11.1 mmol/L)
* Ability to understand and the willingness to sign a written informed consent document.
* Diagnosis from a retinal specialist of ETDRS level of 35 or higher with or without DME or diagnosis from a retinal specialist of ETDRS level 20 or lower and no DME.
* Standard Corrected Visual Acuity of at least 20/40 or better in both eyes.

Exclusion Criteria:

* Currently participating in an interventional eye study (e.g., actively receiving the investigational product for Diabetic Retinopathy (DR) and/or Diabetic Macular Edema (DME)).
* Has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure or glycemic control, microphthalmia, or previous enucleation).
* Pregnancy
* Has a known allergy to or contraindication for the use of Tropicamide 1% or other mydriatic eye drops.
* Any condition that is contraindicated for the use of study devices in the opinion of the investigator.
* Contraindication for imaging by devices used in the study due to any of the following:
* Subject is hypersensitive to light
* Subject recently underwent photodynamic therapy (PDT)
* Subject is taking medication that causes photosensitivity

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 80 eligible subjects, these subjects will be categorized as ETDRS ≥ 35 with or without DME and subjects with ETDRS 20 or less and no DME
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 1 Day
  Agreement of AI device results (mtmDR(+), mtmDR(-)) obtained from fundus cameras

OTHER OUTCOMES:
Exploratory Objective | 1 Day
  Agreement of AI device probability scores obtained from fundus cameras
Exploratory Endpoint | 1 Day
  Agreement of AI device results (mtmDR(+), mtmDR(-), "Exam Quality Insufficient" obtained from fundus cameras

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Singh, BS, Study Director — Digital Diagnostics, Inc.
Locations (1):
- Midwest Eye Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No